CLINICAL TRIAL: NCT04385810
Title: Description of Ophthalmologic Injuries in Intensive Care During the SARS-CoV2 Epidemic - COVID19
Acronym: DOCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JDS_2020_13
Record Dates: First submitted 2020-04-29; First posted 2020-05-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Sars-CoV2
Keywords: ophthalmological lesions
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ophthalmologic exam (Experimental)
  Interventions: Procedure: Ophthalmologic exam

INTERVENTIONS:
Procedure: Ophthalmologic exam — Direct exam and Slit lamp exam Shirmer test Retinophotography At inclusion, day 7, day 14 and discharge from hospital

SUMMARY:
The management of patients with SARS-CoV2 in respiratory distress can expose to corneal or retinal lesions induced by the stay in intensive care.

Examination by ophthalmologists would make it possible to detect the most of the ophthalmologic problems known in intensive care and to provide an early, preventive or curative therapeutic response when possible, in order to avoid irreversible visual loss.

The object of the research is to assess the presence and the importance of surface ophthalmologic lesions, the presence and the importance of retinal or optic nerve lesions, in order to improve the monitoring and primary prevention of this population

ELIGIBILITY:
Inclusion Criteria:

* patient SARS-CoV2 positive (RT-PCR or chest scanner)
* hospitalized in intensive care

Exclusion Criteria:

* traumatic lesion of the face or any other condition preventing any ophthalmological evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Describe ophthalmologic damage to the cornea with direct exam at day 0 | Day 0
  Direct exam
Describe ophthalmologic damage to the cornea with direct exam at day 7 | Day 7
  Direct exam
Describe ophthalmologic damage to the cornea with direct exam at day 14 | Day 14
  Direct exam
Describe ophthalmologic damage to the cornea with direct exam at discharge of hospital | Discharge of hospital, up to 3 months
  Direct exam
Describe ophthalmologic damage to the cornea with slit lamp exam at day 0 | Day 0
  Slit lamp exam
Describe ophthalmologic damage to the cornea with slit lamp exam at day 7 | Day 7
  Slit lamp exam
Describe ophthalmologic damage to the cornea with slit lamp exam at day 14 | Day 14
  Slit lamp exam
Describe ophthalmologic damage to the cornea with slit lamp exam at discharge of hospital | Discharge of hospital, up to 3 months
  Slit lamp exam
Describe tear film anomalies at day 0 | Day 0
  Shirmer test
Describe tear film anomalies at day 7 | Day 7
  Shirmer test
Describe tear film anomalies at day 14 | Day 14
  Shirmer test
Describe tear film anomalies at discharge of hospital | Discharge of hospital, up to 3 months
  Shirmer test
Describe ophthalmologic damage to the retina at day 0 | Day 0
  Retinophotography
Describe ophthalmologic damage to the retina at day 7 | Day 7
  Retinophotography
Describe ophthalmologic damage to the retina at day 14 | Day 14
  Retinophotography
Describe ophthalmologic damage to the retina at discharge of hospital | Discharge of hospital, up to 3 months
  Retinophotography
Describe ophthalmologic damage to the optic nerve at day 0 | Day 0
  Retinophotography
Describe ophthalmologic damage to the optic nerve at day 7 | Day 7
  Retinophotography
Describe ophthalmologic damage to the optic nerve at day 14 | Day 14
  Retinophotography
Describe ophthalmologic damage to the optic nerve at discharge of hospital | Discharge of hospital, up to 3 months
  Retinophotography

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel DEVYS, MD, Principal Investigator — Fondation Adolphe de Rothschild
Locations (1):
- Fondation Adolphe de Rothschild, Paris, France

REFERENCES:
- [Result] Stephan S, Cohen F, Salviat F, Thevenin S, Devys JM, Cochereau I, Gabison E. Evaluation of the impact of intensive care support for COVID-19 on the ocular surface in a prospective cohort of 40 eyes. Ocul Surf. 2021 Oct;22:13-14. doi: 10.1016/j.jtos.2021.06.008. Epub 2021 Jun 23. No abstract available. PMID 34174393